CLINICAL TRIAL: NCT00573690
Title: A Two Arm Phase I Trial of Sorafenib in Combination With Cisplatin/Etoposide or Carboplatin/Pemetrexed in Patients With Solid Tumors
Brief Title: Sorafenib Combined With Cisplatin and Etoposide or Carboplatin and Pemetrexed in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0613; CDR0000579819 (Other: NCI PDQ number); UNC-LCC-07-0971
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Cisplatin; Etoposide; Pemetrexed; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients receive cisplatin IV over 1 hour on day 2 of courses 1 and 2 and on day 1 of all subsequent courses; etoposide IV over 30 minutes on days 1-3; and oral sorafenib tosylate once or twice daily on days 1-21. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: sorafenib tosylate
- Group 2 (Experimental): Patients receive carboplatin IV over 30 minutes and pemetrexed disodium IV over 10 minutes on day 1. Patients also receive sorafenib tosylate as in group 1. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: carboplatin; Drug: pemetrexed disodium; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: carboplatin — Given IV
  Arms: Group 2
Drug: cisplatin — Given IV
  Arms: Group 1
Drug: etoposide — Given IV
  Arms: Group 1
Drug: pemetrexed disodium — Given IV
  Arms: Group 2
Drug: sorafenib tosylate — Given orally

SUMMARY:
RATIONALE: Sorafenib and pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cisplatin, etoposide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with cisplatin and etoposide or carboplatin and pemetrexed may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of sorafenib when given together with cisplatin and etoposide or carboplatin and pemetrexed in treating patients with metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the recommended phase II dose and maximum tolerated dose of sorafenib tosylate when administered in combination with cisplatin and etoposide or carboplatin and pemetrexed disodium in patients with metastatic solid tumors.

Secondary

* To characterize the toxicities of these regimens in these patients.
* To evaluate the efficacy of these regimens in these patients, as measured by RECIST criteria or by tumor markers, if applicable (e.g., PSA, CA-125).
* To determine the pharmacokinetics of sorafenib tosylate when administered in combination with etoposide in these patients (samples are no longer being collected and studies are no longer being performed as of 1/8/09).

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

* Group 1: Patients receive cisplatin IV over 1 hour on day 2 of courses 1 and 2 and on day 1 of all subsequent courses; etoposide IV over 30 minutes on days 1-3; and oral sorafenib tosylate once or twice daily on days 1-21. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.
* Group 2: Patients receive carboplatin IV over 30 minutes and pemetrexed disodium IV over 10 minutes on day 1. Patients also receive sorafenib tosylate as in group 1. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.

Patients in group 1 undergo blood sample collection on day 1 of courses 1 and 2 for pharmacokinetic studies (samples are no longer being collected and studies are no longer being performed as of 1/8/09).

After finishing treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic solid tumor

  * Disease progressed during at least one standard therapy OR has a disease for which there is no standard therapy
* No squamous cell carcinoma of the lung
* Asymptomatic brain metastases allowed provided both of the following criteria are met:

  * Brain metastases were treated ≥ 6 months ago
  * Brain metastases are clinically stable without steroid treatment for 1 week
* No clinically relevant pleural effusions or ascites that cannot be controlled by drainage (group 2)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* INR < 1.5 or PT/PTT normal
* Creatinine clearance ≥ 45 mL/min
* Negative serum pregnancy test
* Fertile patients must use effective contraception during and for at least 2 weeks after completion of study treatment
* No New York Heart Association class III or IV congestive heart failure
* No unstable angina (anginal symptoms at rest) or new onset angina (within the past 3 months)
* No myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension, defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg, despite optimal medical management
* No known severe hypersensitivity to sorafenib tosylate or any its excipients, etoposide, pemetrexed disodium, cisplatin, or carboplatin
* No known HIV infection
* No chronic hepatitis B or C
* No active clinically serious infection > CTCAE grade 2
* No thrombotic or embolic events, such as cerebrovascular accident or transient ischemic attacks, within the past 6 months
* No pulmonary hemorrhage or bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No serious non-healing wound, ulcer, or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy
* No condition that impairs the patient's ability to swallow whole pills
* No malabsorption problem, uncontrolled inflammatory bowel disease, or gastrointestinal disorder causing ≥ 5 bowel movements in a 24-hour period
* No significant traumatic injury within the past 4 weeks
* Able to take vitamin B12 supplementation and folic acid (group 2)

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior major surgery or open biopsy
* No more than 3 prior cytotoxic therapies for metastatic disease
* No concurrent St. John's wort or rifampin
* No non-steroidal anti-inflammatory drugs (NSAIDs) for 2 days before (5 days for long-acting NSAIDs), during, and for 2 days after pemetrexed disodium administration (group 2)
* Concurrent anticoagulation treatment with warfarin or heparin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose and maximum tolerated dose of sorafenib tosylate when administered in combination with cisplatin and etoposide or carboplatin and pemetrexed disodium | 12 months

SECONDARY OUTCOMES:
Toxicity | 12 months
Efficacy of treatment as measured by RECIST criteria or by tumor markers | 36 months
Pharmacokinetics of sorafenib tosylate in combination with etoposide (samples are no longer being collected and studies are no longer being performed as of 1/8/09) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Elizabeth C. Dees, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States